CLINICAL TRIAL: NCT06576843
Title: An Open-label, Multicentre Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Repeated Doses of INDV-6001 in Adults With Moderate to Severe Opioid Use Disorder
Brief Title: INDV-6001 Multiple-Dose Pharmacokinetic Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INDV-6001-201
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Opioid Use Disorder
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination; Sublocade

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): SUBOXONE 12-16 mg once daily (to continue through Day 7), followed by INDV-6001 (600 mg Day 1, followed by 600 mg on Day 8, Day 92, and Day 176)
  Interventions: Drug: INDV-6001; Drug: Suboxone
- Cohort 2 (Experimental): SUBOXONE 12-16 mg once daily (to continue through Day 7), followed by INDV-6001 (600 mg Day 1, followed by 600 mg on Day 8, Day 64, Day 120, and Day 176)
  Interventions: Drug: INDV-6001; Drug: Suboxone
- Cohort 3 (Experimental): SUBOXONE 12-16 mg once daily (to continue through Day 7), followed by INDV-6001 (600 mg Day 1, 600 mg Day 8, followed by 250 mg on Day 15, Day 43, Day 71, and Day 99)
  Interventions: Drug: INDV-6001; Drug: Suboxone
- Cohort 4 (Experimental): SUBOXONE 12-16 mg once daily (to continue through Day 7), followed by INDV-6001 (600 mg Day 1, followed by 100 mg on Day 8, Day 36, Day 64, and Day 92)
  Interventions: Drug: INDV-6001; Drug: Suboxone
- Cohort 1a (Experimental): In Cohort 1, up to 15 participants who reach Day 260 will be enrolled into Cohort 1a. Participants in Cohort 1a will receive an additional injection of INDV-6001 600 mg in the back of the upper arm on Day 260.
  Interventions: Drug: INDV-6001
- Cohort 2a (Experimental): In Cohort 2, up to 15 participants who reach Day 232 will be enrolled into Cohort 2a. Participants in Cohort 2a will receive an additional injection of INDV-6001 600 mg in the thigh on Day 232.
  Interventions: Drug: INDV-6001
- Cohort 3a (Experimental): In Cohort 3, up to 15 participants who reach Day 127 will be enrolled into Cohort 3a. Participants in Cohort 3a will receive an injection of SUBLOCADE 300 mg (abdomen) on Day 127.
  Interventions: Drug: Sublocade
- Cohort 4a (Experimental): In Cohort 4, up to 15 participants who reach Day 120 will be enrolled in Cohort 4a. Participants in Cohort 4a will receive an injection of SUBLOCADE 100 mg (abdomen) on Day 120.
  Interventions: Drug: Sublocade
- Cohort 7 (Experimental): Participants in Cohort 7 who are new to BUP treatment will undergo rapid induction with SUBLOCADE 300 mg (per product labelling) in the abdomen on Day 1 following an initial dose of SUBOXONE (eg, 4 mg).
  All participants in Cohort 7 will receive: SUBLOCADE 300 mg (abdomen) on Day 1 and Day 8, SUBLOCADE 100 mg (abdomen) on Day 36, and 600mg INDV-6001 on Day 64.
  Interventions: Drug: INDV-6001; Drug: Suboxone; Drug: Sublocade

INTERVENTIONS:
Drug: INDV-6001 — Extended-release subcutaneous injection
  Arms: Cohort 1; Cohort 1a; Cohort 2; Cohort 2a; Cohort 3; Cohort 4; Cohort 7
Drug: Suboxone — Oral sublingual film
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 7
Drug: Sublocade — Extended-release subcutaneous injection
  Arms: Cohort 3a; Cohort 4a; Cohort 7

SUMMARY:
This is a multicentre, open-label, multiple dose study of INDV-6001 in adult participants with moderate or severe OUD as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5).

The current study will evaluate the pharmacokinetics (PK), safety, and tolerability of INDV-6001 following multiple doses in participants with OUD to select optimum dosing regimens for future studies. Prior to receiving INDV-6001, participants will be stabilised on 12-16 mg of transmucosal (TM) BUP (SUBOXONE®) or will transition from a 100-mg monthly maintenance dose of SC extended-release BUP (SUBLOCADE®). This study will also evaluate the use of alternative injection sites (thigh, back of upper arm), which may be desirable in this patient population for the anticipated extended durations of treatment.

DETAILED DESCRIPTION:
Study Cohorts:

There are multiple cohorts (1, 2, 3, 4 and 7) testing varying dose strengths and frequencies of INDV-6001 in participants who are not receiving long-acting treatment for OUD. Up to 15 participants from each of the Cohorts 1, 2, 3, and 4 will enrol into Cohorts 1a, 2a, 3a, and 4a, respectively.

Study Periods:

Screening Period: from the Screening Visit until prior to the first SUBOXONE or SUBLOCADE dose as a part of this study Pre-Investigational Medicinal Product (IMP) Period: from the first SUBOXONE or SUBLOCADE dose as a part of this study until prior to the first INDV-6001 dose IMP Period: from the first INDV-6001 dose until the SUBLOCADE injection (Cohorts 3a and 4a only) or until the end of the study (EOS; all remaining cohorts) Post-IMP Period: (Cohorts 3a and 4a only) from the SUBLOCADE injection until EOS

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in any cohort open to enrolment in the study only if all of the following criteria apply:

1. Has signed the ICF and have the ability to understand and comply with the requirements and restrictions listed therein
2. Is an adult (male or female) between the ages of 18 and 65 years, inclusive, at the time of signing the ICF
3. Has a BMI of ≥18.0 to ≤33.0 kg/m2
4. Is seeking MOUD and currently meets or has documented history of moderate or severe OUD as per DSM-5 criteria. For Cohorts 1-4 only: can be dose-adjusted to 12 to 16 mg SUBOXONE QD or currently taking TM BUP for OUD and can be dose-adjusted to 12 to 16 mg SUBOXONE QD
5. Agrees not to take any BUP-containing products, other than those administered for the current study, throughout the duration of the study
6. If a woman of childbearing potential, not pregnant or lactating and agrees to follow contraception guidelines per protocol; if a women of non-childbearing potential (WONCBP), is:

   1. Postmenopausal (defined as no menses for 12 months without an alternative medical cause and confirmed by high FSH level of >30 mIU/mL in women not using hormonal contraception or hormonal replacement therapy) or
   2. Permanently sterilised (eg, bilateral tubal occlusion, bilateral tubal ligation, complete hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
7. If a man, agrees to follow contraception guidelines per protocol 5.2 Exclusion Criteria

A participant will not be eligible for inclusion in this study if any of the following criteria apply:

1. Has current diagnosis or medical condition, other than OUD, requiring chronic opioid treatment
2. Has a concurrent primary substance use disorder, as defined by DSM-5 criteria, other than opioid, tobacco, cannabis, or mild to moderate alcohol use disorders
3. Has an injection area unsuitable for SC injections (eg, nodules, scarring, lesions, excessive pigment) in the areas designated for possible injection in the study
4. Is currently using another MOUD treatment other than TM BUP (eg, SUBOXONE) or has had prior treatment with any long-acting injectable form of a BUP-containing product in the past 18 months (or if 18-24 months with a positive UDS) prior to consent; treatment with oral naltrexone or methadone products within 14 days prior to consent (or positive UDS for methadone at Screening); or treatment with depot naltrexone within the 3 months prior to consent
5. Has had significant traumatic injury or major surgical procedure (as defined by the investigator) within 30 days prior to the first dose of INDV-6001 or still recovering from such prior injury or surgery
6. Has congenital long QT syndrome, history of prolonged QT in the 3 months prior to screening, or a corrected QT interval (Fridericia's - QTcF) >450 msec (male) or >470 msec (female), or history of risk factors for Torsades de Pointes. Has known personal history of taking Class IA antiarrhythmic medications (eg, quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (eg, sotalol, amiodarone) or other mediations that prolong the QT interval
7. Has known family history of congenital QT prolongation or sudden unexplained death
8. Is currently taking (within the 30 days prior to signing the ICF) prescription or OTC medications that are clinically relevant moderate or strong cytochrome P450 (CYP) 3A4 or CYP 2C8 inducers or inhibitors (eg, rifampin, azole antifungals [eg, ketoconazole], macrolide antibiotics [eg, erythromycin])
9. Has a history of suicidal ideation within 30 days prior to providing written informed consent (evidenced by answering yes to either question 1 or 2 on the C-SSRS) or a history of a suicide attempt in the 6 months prior to consent
10. Has any active medical condition (including organ disease), psychiatric illness, social/legal situation (including court order requiring treatment for OUD), or concurrent medication/treatment that may compromise participant safety, interfere with study endpoints, limit compliance with study requirements, or compromise the ability of the participant to provide written informed consent
11. Has active hepatitis B or C as evidenced by positive serology and PCR test confirmation
12. Has total bilirubin ≥1.5 × ULN (with direct bilirubin >20% of total bilirubin), ALT ≥3 × ULN, AST ≥3 × ULN, or INR >1.5 × ULN at Screening)
13. Has serum creatinine >1.5 × ULN or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 by CKD-EPI formula
14. Has known allergy or hypersensitivity to BUP, any excipients of INDV-6001, SUBOXONE, or SUBLOCADE
15. Is currently participating in another interventional clinical study, and/or has been treated with investigational product INDV-2000 within 1 month prior to Screening Visit, or another investigational agent within 3 months prior to Screening Visit
16. Is currently being treated with medications contraindicated for use with BUP as per local prescribing information
17. Has donated more than 500 mL of blood within the past 3 months prior to consent
18. Is a member of site staff, has a financial interest in Indivior, or is an immediate family member of anyone directly involved in the study (eg, site staff or Indivior employee)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  AUCtau for Cohorts 1-4
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  Cmax for Cohorts 1-4
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  Tmax for Cohorts 1-4
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  Cmin for Cohorts 1-4
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  Ctrough for Cohorts 1-4
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 injection in the abdomen | Up to 260 days
  Cavg for Cohorts 1-4
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 injection | Up to 260 days
  % fluctuation for Cohorts 1-4
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  AUCtau for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  Cmax for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  Tmax for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  Cmin for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  Ctrough for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  Cavg for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 injection in the back of the upper arm Vs abdomen injection location | Up to 168 days [24 weeks]
  % fluctuation for Cohort 1a [Day 260 injection in the back of the upper arm] Vs Cohort 1 [Day 176 Injection in the abdomen]
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  AUCtau for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  Cmax for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  Tmax for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  Cmin for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  Ctrough for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  Cavg for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 injection in the Thigh Vs abdomen injection location | Up to 128 days [16 weeks]
  % fluctuation for Cohort 2a [Day 232 injection in the Thigh] Vs Cohort 2 [Day 176 injection in the abdomen]

SECONDARY OUTCOMES:
Assessment of the safety and tolerability of INDV-6001 injection | Up to 260 days
  Incidence, severity, and relatedness of treatment-emergent adverse events (TEAEs), serious TEAEs, TEAEs leading to discontinuation, fatal TEAEs, and AEs of special interest (AESIs) for All Cohorts
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  AUCtau for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  Cmax for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  Tmax for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  Cmin for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  Ctrough for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  Cavg for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 250mg injection in the abdomen Vs SUBLOCADE 300mg injection in the abdomen | Up to 56 days [8 weeks]
  %fluctuation for Cohort 3 [Day 99 250mg INDV-6001 injection in the abdomen] Vs Cohort 3a [Day 127 300mg SUBLOCADE injection in the abdomen]
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  AUCtau for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  Cmax for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  Tmax for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  Cmin for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  Ctrough for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  Cavg for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 100mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 56 days [8 weeks]
  % fluctuation for Cohort 4 [Day 92 250mg INDV-6001 injection in the abdomen] Vs Cohort 4a [Day 120 100mg SUBLOCADE injection in the abdomen]
Steady-state area under the plasma concentration-time curve over the dosing interval (AUCtau) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  AUCtau for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state maximum observed plasma concentration (Cmax) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  Cmax for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state time to attain the maximum observed plasma concentration (Tmax) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  Tmax for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state minimum plasma concentration over a dosing interval (Cmin) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  Cmin for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state plasma concentration measured at the end of the dosing interval (Ctrough) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  Ctrough for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state average plasma concentration over the dosing interval (Cavg) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  Cavg for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]
Steady-state ratio of peak to trough plasma concentrations over a dosing interval (% fluctuation) of buprenorphine following INDV-6001 600mg injection in the abdomen Vs SUBLOCADE 100mg injection in the abdomen | Up to 112 days [16 weeks]
  % fluctuation for Cohort 7 [Day 64 600mg INDV-6001 injection in the abdomen] Vs [Day 36 100mg SUBLOCADE injection in the abdomen]

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Artemis Institute for Clinical Research, San Diego, California
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Precise Research Centers, Flowood, Mississippi
  - Hassman Research Institute (Cenexel HRI - Marlton), Marlton, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research, Dayton, Ohio
  - Insite Clinical Research, LLC, DeSoto, Texas
  - Memorial Hermann Village, Houston, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Progressive Clinical Research, Bountiful, Utah